CLINICAL TRIAL: NCT06336278
Title: The Relationship Between Central Sensitization and Kinesiophobia in Patients With Knee Osteoarthritis
Brief Title: Relationship Between Central Sensitization and Kinesiophobia in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Selda Sarıkaya (Other)
Responsible Party: Sponsor-Investigator, Selda Sarıkaya, Principal Investigator, Clinical Professor, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Other Study IDs: 19/03/2024
Record Dates: First submitted 2024-03-19; First posted 2024-03-28 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis; Central Sensitisation; Kinesiophobia
Keywords: pain pressure treshold; algometer; knee osteoarthritis; central sensitization; kinesiophobia
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee Osteoarthritis: Patients who have knee pain at least 6 months, 45-75 years old, kellgren-lawrence grade 1-3
  Interventions: Diagnostic Test: Pressure Algometer
- Control: Subjects who have not knee pain, 45-75 years old
  Interventions: Diagnostic Test: Pressure Algometer

INTERVENTIONS:
Diagnostic Test: Pressure Algometer — Pressure algometer is used to detect pain pressure treshold.

SUMMARY:
Objective: The knee joint is one of most common locations in OA. In recent years, it has been accepted that there are different pain phenotypes and patient subgroups in knee OA and that central sensitization (CS) mechanisms are at the forefront in some patients. It is also known that fear of movement, known as kinesiophobia, develops in patients with chronic pain. The aim of this study is to investigate CS and kinesiophobia in patients with knee OA, their relationships with each other, and their effects on pain intensity, functional status, pain catastrophizing and depression.

Materials and Methods: Forty-two patients with knee OA and 42 healthy subjects participated in our study. Demographic data, body mass index, habits, comorbidities, medications of participants and disease duration and radiographic grade of knee OA patients were recorded. VAS was used to assess the severity of pain and WOMAC was used to assess pain and functional status in patients with OA. Algometer (pressure pain threshold measurement) and Central Sensitization Inventory were used to evaluate central sensitization in all participants. Pressure pain threshold (PPT) was measured at 3 different points: knee joint, cruris and forearm. The presence of kinesiophobia was assessed with the Tampa Scale af Kinesiophobia (TSK). Pain Catastrophizing Scale (PCS) and Beck Depression Inventory (BDI) were used to assess chronic pain related symptoms.

DETAILED DESCRIPTION:
Forty-two patients with knee OA and 42 healthy subjects participated in our study. Demographic data, body mass index, habits, comorbidities, medications of participants and disease duration and radiographic grade of knee OA patients were recorded. VAS was used to assess the severity of pain and WOMAC was used to assess pain and functional status in patients with OA. Algometer (pressure pain threshold measurement) and Central Sensitization Inventory were used to evaluate central sensitization in all participants. Pressure pain threshold (PPT) was measured at 3 different points: knee joint, cruris and forearm. The presence of kinesiophobia was assessed with the Tampa Scale af Kinesiophobia (TSK). Pain Catastrophizing Scale (PCS) and Beck Depression Inventory (BDI) were used to assess chronic pain related symptoms.

ELIGIBILITY:
Inclusion Criteria for knee osteoarthritis group:

* Being a healthy volunteer between the ages of 45-75
* Being diagnosed with knee osteoarthritis according to ACR diagnostic criteria
* Knee pain for at least 6 months
* Kellgren-Lawrence 1, 2 or 3 radiologic grade of knee OA
* Body mass index below 35

Exclusion Criteria for knee osteoarthritis group:

* Presence of chronic widespread painful diseases other than osteoarthritis (fibromyalgia syndrome etc.), rheumatologic disease, peripheral neuropathy
* Presence of uncontrolled systemic disease
* Cooperation limitation or cognitive impairment
* Active arthritis in the knee joint to be evaluated
* Presence of prosthesis in the knees
* Pain in the forearm
* Body mass index of 35 and above

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria for control group:
  * Being a healthy volunteer between the ages of 45-75
  * No pain in the knee and forearm
  * No mechanical, inflammatory, endocrine, degenerative, degenerative, systemic comorbidities that may affect the knee joint
  * Body mass index below 35
  Exclusion Criteria for control group:
  * Diagnosed with knee osteoarthritis
  * Presence of uncontrolled systemic disease
  * Cooperation limitation or cognitive impairment
  * Presence of chronic painful disease, rheumatologic disease, peripheral neuropathy
  * Body mass index of 35 and above
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Treshold | Day 1
  Algometer was used to detect pressure pain threshold. Higher scores mean better outcomes.
Central Sensitization | Day 1
  Central Sensitization Inventory was used to evaluate central sensitization. Minimum value is 0 , maximum value is 100. Higher values means worse outcomes.
Kinesiophobia | Day 1
  The presence of kinesiophobia was assessed with Tampa Scale af Kinesiophobia. Minimum value is 17 , maximum value is 68. Higher values means worse outcomes.

SECONDARY OUTCOMES:
Pain Catastrophizing | Day 1
  Pain Catastrophizing Scale was used to assess chronic pain related symptoms. Minimum value is 0 , maximum value is 52. Higher values means worse outcomes.
Depression | Day 1
  Beck Depression Inventory was used to assess depression. Minimum value is 0 , maximum value is 63. Higher values means worse outcomes.
Visuel Analog Scala | Day 1
  Visuel Analog Scala was used to assess pain intensity. Patients' pain (0=no pain, 10=intolerable pain) on a 100 mm horizontal line. The marked value was recorded in millimeters.
Western Ontario and McMaster Universitesies Osteoarthritis Index | Day 1
  Pain and functional status of the patients included in our study assessment was performed using this index, consists of a total of three subscales and 24 questions, each question is scored between 0 and 4 (0=none, 4=very severe). Minimum value is 0, maximum value is 100. Higher scores indicate an increase in pain and stiffness and a decline in physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit Universitiy, Zonguldak, Turkey (Türkiye)